CLINICAL TRIAL: NCT06216470
Title: Phase II Investigator-Initiated Study to Understand the Vaccinal Effect of HBsAg Monoclonal Ab VIR-3434 in Chronic Hepatitis B Infection
Brief Title: Vaccinal Effect of HBsAg Monoclonal Ab VIR-3434 in Chronic Hepatitis B Infection [VISION]
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-5492
Record Dates: First submitted 2024-01-08; First posted 2024-01-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- VIR-3434 (Experimental): VIR-3434 300 mg subcutaneous injection every 4 weeks*48 weeks
  Interventions: Drug: VIR-3434

INTERVENTIONS:
Drug: VIR-3434 — VIR-3434 is a human monoclonal antibody that binds the antigenic loop present in all forms of the surface envelope protein (small, middle, and large HBsAg).

SUMMARY:
This is a Phase II Investigator-Initiated Study to understand the vaccinal effect of HBsAg monoclonal Ab VIR-3434 in chronic hepatitis B infection.

The purpose of this study is to test VIR-3434, an experimental drug that specifically targets the HBsAg of hepatitis B virus, to clear it from the body.

This is an open label study and there is no placebo used in this study. All participants will receive the VIR-3434 for 48 weeks and then follow up in the study for 48 weeks. A total duration of approximately 104 weeks including screening period for the entire study.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the vaccinal effect of VIR-3434 in chronic HBeAg-negative hepatitis B (CHB) patients suppressed on nucleos(t)ide analogue therapy. Total 15 patients will be enrolled at single site.

The participants will receive VIR-3434 300 mg subcutaneous injection every 4 weeks x 48 weeks and then follow up for 48 weeks. Total three Fine-needle aspiration (FNA) procedure will be performed during the study: before treatment, 3 days after the first injection and 3 days after the week24 injection.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 to ≤65 years
2. Chronic HBV infection with evidence of HBsAg-positivity x > 6 months
3. Quantitative HBsAg 300 - 10,000 IU/mL
4. On stable nucleos(t)ide therapy >1 year
5. HBV DNA < 60 IU/mL on 2 occasions at least 12 weeks apart
6. ALT ≤ 45 U/L on 2 occasions at least 12 weeks apart
7. Female subjects must have a negative pregnancy test or confirmation of postmenopausal status. Women of child-bearing potential (WOCBP) must have a negative pregnancy test at screening and on Day 1, cannot be breast feeding, and must be willing to use highly effective methods of contraception 14 days before study drug administration through the study participation. Female subjects must also agree to refrain from egg donation and in vitro fertilization from the time of study drug administration through the study participation.
8. Male subjects with female partners of child-bearing potential must agree to meet 1 of the following contraception requirements from the time of study drug administration through the study participation: documentation of vasectomy or azoospermia, or male condom use plus partner use of 1 of the contraceptive options listed for contraception for WOCBP. Male subjects must also agree to not donate sperm from the time of study drug administration through the study participation.
9. Able and willing to sign informed consent

Exclusion Criteria:

1. History of cirrhosis as evidenced by prior Liver Elastography (Fibroscan) > 12 kilopascals (kPa), liver biopsy (F4 by METAVIR) or clinical evidence of decompensation (ascites, hepatic encephalopathy)
2. History of or current hepatocellular carcinoma
3. Hepatitis C Virus (HCV) RNA or anti-Hepatitis D Virus (HDV) positive
4. HIV co-infection
5. Pregnancy or lactation
6. Alanine Aminotransferase (ALT) > 45 U/L
7. History of chronic liver disease other than HBV aside from fatty liver documented only on US
8. Use of peginterferon therapy for HBV infection within past 12 months
9. Use of chronic immunosuppressive medications at a dose equivalent to 10 mg daily of prednisone or greater within past 6 months
10. Other significant medical illness that might interfere with this study: significant pulmonary dysfunction in previous 6 months, malignancy other than non-melanoma skin cancer in previous 5 years, immunodeficiency syndrome
11. Subject has received any investigational drug (including any investigational vaccines) within 90 days or 5 half-lives (whatever is longer) before screening for this study or is currently enrolled in an investigational study
12. Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments, such as liver FNAs
13. Platelet count < 120,000,000,000/L
14. The International Normalised Ratio (INR) > 1.3
15. Bilirubin > 40 µmol/L
16. Hemoglobin < 110 g/dL for women or 120 g/dL for men
17. estimated Glomerular Filtration Rate (eGFR) < 45 cc/min
18. Alpha Fetoprotein (AFP) > 50 ng/mL
19. Prior liver or other solid organ transplantation
20. Patients on anticoagulation therapy or with any bleeding diathesis
21. Patients with hemoglobinopathy (thalassemia, sickle cell disease etc)
22. Other significant liver disease: alcoholic liver disease, autoimmune hepatitis, hemochromatosis, primary biliary cholangitis, primary sclerosing cholangitis, Wilson Disease or alpha-1 antitrypsin deficiency - as documented in clinical history
23. Unable to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in log Quantitative HBsAg | from baseline through study completion, an average of 2 year

SECONDARY OUTCOMES:
Absolute and change of Hepatitis B Virus (HBV) RNA | from baseline through study completion, an average of 2 year
Absolute and change of HBV core-related Ag | from baseline through study completion, an average of 2 year
Proportion of subjects with HBsAg loss | from baseline through study completion, an average of 2 year
HBeAg seroconversion | from baseline through study completion, an average of 2 year
  Proportion of subject with HBeAg seroconversion
Frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) with study treatment | from baseline through study completion, an average of 2 year
  Frequency of AEs and SAEs with VIR-3434 administration in combination with NA therapy for CHB
Frequency of AEs and SAEs due to hepatic FNA | from baseline through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Feld, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No